CLINICAL TRIAL: NCT00510198
Title: PRECEDE-HF -Prospective, Randomized Evaluation of Cardiac Compass With OptiVol in the Early Detection of Decompensation Events for Heart Failure
Brief Title: Evaluation of Cardiac Compass With OptiVol in the Early Detection of Decompensation Events for Heart Failure
Acronym: PRECEDE-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study enrollment significantly below protocol expectation
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 603
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-03

CONDITIONS: Congestive Heart Failure
Keywords: Heart Disease; Congestive Heart Failure; Thoracic Fluid Monitoring
MeSH Terms: conditions — Heart Failure; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm 1: SOC and CC with OptiVol (Active Comparator): Standard of Care and Cardiac Compass with OptiVol as the Control. Intervention is standard of care, such as symptom assessment with the addition of viewing Cardiac Compass trends and the OptiVol diagnostic.
  Interventions: Device: Cardiac Compass with OptiVol Fluid Status Monitoring
- Control Arm 2: SOC (Active Comparator): Intervention is Standard of Care alone, such as assessment of symptoms, only. Device trending information, but OptiVol is not allowed.
  Interventions: Device: Standard of Care alone (clinical assessment)

INTERVENTIONS:
Device: Cardiac Compass with OptiVol Fluid Status Monitoring — Review of Cardiac Compass with OptiVol Fluid Status Monitoring
  Arms: Control Arm 1: SOC and CC with OptiVol
Device: Standard of Care alone (clinical assessment) — Clinical assessment utilizing standard of care, alone.
  Arms: Control Arm 2: SOC

SUMMARY:
The purpose of the PRECEDE-HF study is to collect data to compare patients whose heart failure is managed using Cardiac Compass with OptiVol (which is a tool in the device that records information about the heart that doctors can use to help treat their heart disease) combined with standard treatment methods (Access Group) to patients whose heart failure is managed by standard treatment methods only (Control Group). This comparison will show if the additional monitoring provided by Cardiac Compass with OptiVol delays the time patients are first admitted to hospital for heart failure or delays the time to death.

DETAILED DESCRIPTION:
PRECEDE-HF was a prospective, multi-center, randomized, investigational device exemption (IDE) clinical study. The purpose of this study was to collect data required to determine whether the use of Cardiac Compass including OptiVol Fluid Status Monitoring with standard clinical assessment ("Access Arm") will result in a longer time to first heart failure hospitalization or death compared to standard clinical assessment alone ("Control Arm") and to support the approval of the following device features:

* OptiVol Alert (audible and home monitor alerts) for use in Medtronic devices
* SentryCheck™ Monitor
* OptiVol Alert Suspend (OptiVol enhancement)
* OptiVol Reference Impedance Adjustment (OptiVol enhancement)

ELIGIBILITY:
Inclusion Criteria

The following criteria apply to all subjects:

* Subject has a CRT-D or dual chamber ICD with Cardiac Compass and OptiVol Fluid Status Monitoring implanted in the pectoral region at least 30 days prior to enrollment. CRT-D/ICD must be supported by the Medtronic CareLink Network.
* Subject has a market-released, transvenous, high voltage RV lead
* Subject has a market-released RA lead
* If subject has an LV lead, it must be compatible, not Y-adapted and not currently under investigation
* Subject's heart failure regimen (i.e. beta blocker and ACE inhibitor (or substitute) unless documented evidence of intolerance is available) adheres to current ACC/AHA guidelines for management of chronic heart failure in adult patients
* Subject has a history of at least one heart failure related hospitalization, Emergency Department (ED) visit, or urgent visit necessitating IV diuretic, IV inotropic, IV vasodilator, or other parenteral therapy within 12 months prior to baseline evaluation
* Subject is at least 18 years of age
* Subject is willing and able to comply with the Clinical Investigation Plan (e.g. willing and able to remain available for follow-up visits, use SentryCheck, etc.)
* Subject is willing and able to transmit data using the Medtronic CareLink Network
* Subject (or subject's legally authorized representative) is willing and able to sign and date the study Informed Consent and HIPAA Authorization (U.S.)

Exclusion Criteria

The following criteria apply to all subjects:

* Subject is post heart transplant or actively listed on the transplant list and reasonable probability (as defined by investigator) of undergoing transplantation in the next year
* Subject received a coronary artery bypass graft or valve surgery in the last 90 days
* Subject had a myocardial infarction (MI) in the last 90 days.
* Subject is indicated for valve replacement/repair
* Subject's life expectancy due to non-cardiac reasons is less than six months
* Subject has serum creatinine > 2.5 mg/dL measured within 30 days prior to enrollment.
* Subject is on chronic renal dialysis
* Subject is on continuous or intermittent (> 2 stable infusions per week) infusion therapy for HF
* Subject has complex and uncorrected congenital heart disease
* Subject is enrolled in a Disease Management Program where an outside vendor, company or service is employed to determine, monitor, and/ or alert a clinician or subject to weight changes or other HF signs or symptoms via interactive or passive systems
* Subject is implanted with a cardiac hemodynamic monitor or left ventricular assist device(LVAD)
* Subject is enrolled in a concurrent study, with the exception of a study approved by the Medtronic PRECEDE-HF Clinical Trial Leader prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PRECEDE-HF Study Team, Study Chair — Medtronic
Locations (33):
- United States (33):
  - Anchorage, Alaska
  - Little Rock, Arkansas
  - Berkeley, California
  - Larkspur, California
  - Colorado Springs, Colorado
  - Fort Collins, Colorado
  - Jacksonville, Florida
  - Atlanta, Georgia
  - Kankakee, Illinois
  - Oak Lawn, Illinois
  - Rockford, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Takoma Park, Maryland
  - Springfield, Massachusetts
  - Saginaw, Michigan
  - Ypsilanti, Michigan
  - Saint Cloud, Minnesota
  - Saint Joseph, Missouri
  - St Louis, Missouri
  - Albany, New York
  - Akron, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Elyria, Ohio
  - Oklahoma City, Oklahoma
  - Doylestown, Pennsylvania
  - Lancaster, Pennsylvania
  - Nashville, Tennessee
  - Austin, Texas
  - Richmond, Virginia
  - Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 120 subjects were enrolled but 3 were not randomized into the study for not meeting the inclusion/exclusion criteria.
Groups:
- Access Arm: Standard of Care and Cardiac Compass with OptiVol
- Control Arm: Standard of Care alone
Period: Overall Study
Arm/Group | Access Arm | Control Arm
Started (3 subjects were exited prior to randomization for not meeting the inclusion /exclusion criteria.) | 59 | 58
Completed | 54 | 54
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Access Arm | Control Arm | Total
Number analyzed (Participants) | 59 | 58 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 23 | 44
  >=65 years | 38 | 35 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (17.3) | 63.8 (15.1) | 64.7 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 23 | 36
  Male | 46 | 35 | 81
Region of Enrollment [Number; unit: participants]
  United States | 59 | 58 | 117

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Heart-Failure Hospitalization or All-Cause Death
Description: A composite endpoint of heart-failure hospitalization or all-cause death. To demonstrate a longer time to first heart failure (HF) hospitalization or death in HF subjects managed with standard clinical assessment using Cardiac Compass Trends with OptiVol Fluid Status Monitoring ("Access Arm") compared to HF subjects managed with standard clinical assessment alone ("Control Arm")
Time Frame: Up to five years
Population: all randomized subjects; intention to treat
Measure: Number; unit: Participants with an Event
Arm/Group | Access Arm | Control Arm
Number analyzed (Participants) | 59 | 58
Participants with an Event | 14 | 9
Statistical Analysis 1: Comparison: Access Arm vs Control Arm; This is a log-rank test, which uses the time from randomization to first composite endpoint event to compare the risk of event between Access and Control arms; Test type: Superiority or Other; p = 0.23, Log Rank — The log-rank test was conducted at an alpha level of 0.05. The study was terminated early due to enrollment significantly below protocol expectation. Due to the low sample size and consequently low statistical power, no conclusion can be drawn

2. Primary Outcome: Number of Subjects Proportion Who Have a Safety Composite Event Within the First 6 Months Post-randomization Between the Access Arm and the Control Arm
Description: A safety composite event is defined as an event that includes one or more of the following: Syncope, Worsening renal function resulting in IV therapy, ultrafiltration, or dialysis, Hypotension and/or hypovolemia resulting in the administration of IV fluids, Clinically significant electrolyte abnormalities resulting in IV replacement or ER/hospitalization for correction, Appropriately detected sustained VT/VF episode, Death
Time Frame: Up to five years
Population: all randomized subjects; intention to treat
Measure: Number; unit: Number of Participants with a Event
Arm/Group | Access Arm | Control Arm
Number analyzed (Participants) | 59 | 58
Number of Participants with a Event | 16 | 13
Statistical Analysis 1: Comparison: Access Arm vs Control Arm; Test type: Non-Inferiority or Equivalence — Pre-specified non-inferiority margin was 7.5%; p = 0.36, Two-sample test of proportions — The study was terminated early due to enrollment significantly below protocol expectation. Due to the low sample size and consequently low statistical power, no conclusion can be drawn; Risk Difference (RD) = 4.7, 95% CI 2-sided [-10.9 to 20.3] — The risk difference estimate is the difference between the Access Arm and Control arm

3. Secondary Outcome: Combined Endpoint of All-cause Mortality and Cardiovascular Hospitalizations
Description: To demonstrate a reduction in the combined endpoint of all-cause mortality and cardiovascular hospitalizations in the Access Arm compared to the Control Arm
Time Frame: up to five years
Population: Study was stopped early, therefore secondary objectives were not analyzed.
Groups:
- Access Arm: Standard of Care and Cardiac Compass With OptiVol: Standard of Care and Cardiac Compass with OptiVol
  Cardiac Compass with OptiVol Fluid Status Monitoring: Review of Cardiac Compass with OptiVol Fluid Status Monitoring
- Control Arm: Standard of Care Alone: Standard of Care alone
  Standard of Care alone (clinical assessment): Clinical assessment utilizing standard of care, alone.
Arm/Group | Access Arm: Standard of Care and Cardiac Compass With OptiVol | Control Arm: Standard of Care Alone
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Cardiovascular Hospitalizations
Description: To demonstrate a reduction in cardiovascular hospitalizations in the Access Arm compared to the Control Arm
Time Frame: up to five years
Population: The study was stopped early, therefore secondary objectives were not able to be analyzed.
Arm/Group | Access Arm: Standard of Care and Cardiac Compass With OptiVol | Control Arm: Standard of Care Alone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to five years
Description: Definition of Serious AE: Any significant adverse experience, including those which may be either life threatening or involve permanent or long term injuries, but excluding injuries that are non-life threatening and that are temporary and reasonably reversible.
Arm/Group | Access Arm | Control Arm
Serious Adverse Events (participants affected / at risk) | 32/59 | 21/58
Other Adverse Events (participants affected / at risk) | 11/59 | 3/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Access Arm (N=59) | Control Arm (N=58)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1)
ACUTE DECOMPENSATED HEART FAILURE (Cardiac disorders) | 17 (40) | 11 (31)
ANEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 2 (2) | 1 (1)
ASCITES (General disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CAROTID ARTERY STENOSIS (Vascular disorders) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 1 (1) | 0 (0)
CENTRAL LINE INFECTION (Infections and infestations) | 1 (1) | 1 (1)
CHEST PAIN (Cardiac disorders) | 1 (1) | 0 (0)
CHEST PAIN (NON-CARDIAC) (General disorders) | 0 (0) | 1 (1)
CHOLECYSTECTOMY (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
CIRROHSIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DIGOXIN TOXICITY (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
DRUG INTOLERANCE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
DYSPNEA (Cardiac disorders) | 1 (1) | 1 (1)
EDEMATOUS WEIGHT GAIN (Cardiac disorders) | 1 (1) | 0 (0)
FOOT ULCER (Endocrine disorders) | 0 (0) | 1 (1)
FOREIGN BODY IN GI TRACT (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROENTERITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GERD (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI BLEED (Gastrointestinal disorders) | 0 (0) | 1 (1)
GOUT (Immune system disorders) | 1 (1) | 0 (0)
HYPOTENSION (Cardiac disorders) | 1 (1) | 1 (1)
IMPLANT SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
INJURY TO HAND NOS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ISCHEMIC HEART DISEASE (Cardiac disorders) | 0 (0) | 1 (1)
LEAD CONDUCTOR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LUMBAR VERTEBRAL FRACTURE L1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NEAR SYNCOPE (Cardiac disorders) | 1 (1) | 0 (0)
OVERSENSING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PARALYTIC ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
PYELONEPHRITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
RECTAL PROLAPSE (Gastrointestinal disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 4 (4) | 4 (4)
RENAL INSUFFICIENCY (Renal and urinary disorders) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 2 (2)
SYNCOPE (Cardiac disorders) | 1 (1) | 1 (1)
THYROID MASS (Endocrine disorders) | 0 (0) | 1 (1)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Access Arm (N=59) | Control Arm (N=58)
ACUTE DECOMPENSATED HEART FAILURE (Cardiac disorders) | 4 (4) | 0 (0)
ANXIETY (Psychiatric disorders) | 3 (3) | 1 (1)
GOUT (Immune system disorders) | 4 (6) | 2 (2)

LIMITATIONS AND CAVEATS:
Because none of primary objectives of the study have been met, the pre-specified analyses for all secondary objectives were not performed (per study protocol).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No